CLINICAL TRIAL: NCT07383753
Title: Virtual Hand-Arm Assessments for Children With Cerebral Palsy: Helping Us to Achieve Equity in Rehabilitation Care and Research
Brief Title: Virtual Assessments
Status: Recruiting | Type: Observational
Sponsor: Holland Bloorview Kids Rehabilitation Hospital (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Elaine Biddiss, Principal Investigator, Holland Bloorview Kids Rehabilitation Hospital
Other Study IDs: 4171
Record Dates: First submitted 2025-12-09; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Cerebral Palsy (CP); Developmental Disability; Pediatric Motor Disorders; Motor Skills Disorders
Keywords: Virtual assessment; Tele-rehabilitation; Remote upper limb assessment; Virtual care; Pediatric rehabilitation
MeSH Terms: conditions — Cerebral Palsy; Developmental Disabilities; Motor Skills Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children with Cerebral Palsy (CP): children and adolescents aged 6 to 17 years with a confirmed diagnosis of cerebral palsy and functional hand-arm abilities classified within MACS Levels I-III. All participants must have the cognitive and physical capacity to participate in virtual assessments lasting up to 30 minutes at a time, access to a device and internet connection suitable for videoconferencing, and a caregiver willing to participate in study procedures and provide input on preferences and experiences. Participants complete a standardized series of virtual and in-person upper-limb assessments, wear wrist-worn inertial sensors at home for five days, and contribute caregiver- and child-reported feedback on feasibility, acceptability, and preferences.
  Interventions: Other: Upper-Limb Virtual and In-Person Assessment

INTERVENTIONS:
Other: Upper-Limb Virtual and In-Person Assessment — Participants complete a standardized upper-limb assessment protocol that includes two virtual videoconference assessments-delivered one week apart to evaluate test-retest reliability-and one in-person clinic assessment with the same research therapist to enable within-participant comparison of virtual and in-person scores. After each session, children, caregivers, and therapists complete brief surveys assessing feasibility, ease of completion, acceptability, and preferences.
  Participants also wear bilateral wrist-worn inertial sensors for five consecutive days at home to collect continuous data on naturalistic upper-limb activity. Families also provide caregiver-recorded videos of the child performing two preselected meaningful activities in their home environment. These videos are later scored using the Perceived Quality Rating Scale (PQRS) to evaluate individualized functional performance.

SUMMARY:
Cerebral palsy (CP) affects approximately 1 in 500 Canadian children, and the majority experience hand and arm limitations that impact independence, participation in daily activities, and overall quality of life. Many children require ongoing clinical assessments and therapy delivered in specialized centres, creating significant burden related to travel, scheduling, and interruptions to school and work. Barriers such as geography, socioeconomic factors, and pandemic-related service disruptions have further limited equitable access to in-person care. Although virtual care has expanded rapidly and families have expressed strong interest in hybrid care models, there is currently no validated approach for conducting comprehensive virtual hand-arm assessments for children with CP. Virtual administration of standardized assessments, individualized goal-based evaluations, and naturalistic observation tools has not been systematically studied. Evidence is urgently needed to determine which assessments can be administered virtually, how acceptable and feasible they are for families, and whether virtual and in-person assessment methods produce equivalent results.

DETAILED DESCRIPTION:
Cerebral Palsy (CP) impacts 1 in 500 Canadian children and most (60-83%) have hand/arm limitations that adversely affect independence in daily activities, school, leisure, and social participation. Optimizing hand/arm abilities via therapeutic, surgical and pharmaceutical interventions is a key focus of CP management for children, parents, and clinicians and can involve many clinic appointments for assessments, therapeutic interventions, and follow-up. At best, this introduces a significant family burden with children missing school and potentially other extra-curricular activities and parents juggling work, scheduling and costs. At worst, it means that many children with CP do not receive rehabilitation services and are systemically underrepresented in clinical research studies that could positively impact their lives. Barriers to in-person care include geographic considerations, time/scheduling, availability, socioeconomic factors, not to mention COVID-19-related interruptions. One potential solution to promote equitable and family-focused access to care is to grow capacity for virtual care that can be managed remotely (e.g. via phone/video).

There is a growing movement "not to return to normal" post-COVID, but rather to use the technological advances and learnings to "expand the range, nature and locations of our services for children with developmental disabilities and their families." Many organizations, including our knowledge partner Holland Bloorview Kids Rehabilitation Hospital (HB), have committed to continuing and expanding virtual care options in response to positive family feedback that supports hybrid (virtual/in-person) models of care. This research priority is shared by the wider community of pediatric rehabilitation. Importantly, the goal is not to displace in-person care; rather it is to understand when virtual options can and cannot be offered. It is essential that virtual care, like in-person care, be evidence-based and aligned with current best research findings, clinical expertise and patient/client preferences.

While novel ways of delivering hand-arm therapy via videoconferencing and caregiver engagement have been innovated, it is still difficult to assess hand-arm skills virtually. Hand-arm rehabilitation must be guided by reliable assessment via a combination of patient-reported outcome measures (PROMs), direct measurement, and therapist observations to capture the function, activity, and participation domains of the World Health Organization's International Classification of Function, Disability, and Health (WHO ICF). Outside of PROMs, there are no validated tools for virtual hand-arm assessment of children with CP. This project will focus on direct- and therapist-observed tools to complement digitally-based PROMs that are already suitable for use in virtual assessment. It will address critical issues in need of systematic research as identified in the literature, specifically: What hand-arm assessments can be done virtually? And, what do families want and need in virtual assessments? This study aims to validate well-established standardized measures for virtual administration to support current research and clinical practice, while also exploring individualized measures that can capture the child engaging in their own environment. The ability to observe children in their natural context is seen as an added advantage of virtual assessment.

This critical and timely work is needed to ensure continuation/expansion of the positive practice changes made to overcome access-to-care barriers. Promoting equity, diversity and inclusion in the healthcare system is an urgent priority of health agencies across Canada. Advancing virtual assessment is a complementary and foundational step towards research and practice of evidence-based virtual interventions. This research will quickly generate evidence on the use of existing tools for virtual assessment and what is achievable in the home context. It will contribute new learnings on assessments that can capture the child more naturally in their own environment. This study will identify areas where virtual assessment may not be advisable with currently available tools and provide family-directed learnings for future work.

This study will adopt a convergent mixed methods design including a test-retest approach to compare the feasibility, acceptability, and equivalence of virtual and in-person hand/arm assessments. 100 children and their caregivers will complete the 1 - 1.5 hour assessment protocol twice, once in clinic and once virtually at home via Zoom video-conferencing. A therapist will oversee both assessments. The virtual assessment will occur first. One week later, families will do a second virtual assessment with the same therapist to establish test-retest reliability and to capture any changes in their experience of or perspectives on virtual assessments. The virtual assessment will occur 1 - 3 days after the re-test. Feasibility, acceptability, and equivalence of in-person and virtual assessment will be investigated through quantitative and qualitative methods. For the latter, this study will purposefully recruit (i.e. with diversity as a focus) 25 parents and 25 children for follow-up interviews. All 6 research therapists will also be interviewed after their final session on the risks, opportunities and challenges of virtual assessment.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of Cerebral Palsy
* Are between 6 to 17 years old with sufficient cognitive capacity and cooperation to sit without a break for 30 minutes at a time
* MACS levels I (handles objects easily) to III (handles objects with difficulty)
* No visual limitations that would interfere with video conferencing
* Has a caregiver willing to participate and can questions about preferences
* Have an appropriate device and internet access for video conferencing

Exclusion Criteria:

- Active treatments (e.g. Botulinum Toxin injections or constraint therapy in the last two months, or upper extremity surgery in the last 6 months) that might impact upper limb function stability over the study period.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study population consists of children and adolescents aged 6 to 17 years with a confirmed diagnosis of cerebral palsy who have functional hand and arm abilities classified within Manual Ability Classification System (MACS) Levels I-III. Participants must have sufficient cognitive and physical capacity to participate in virtual videoconference-based assessments for up to 30 minutes at a time and must have access to an internet-enabled device suitable for completing virtual sessions. Each participant must be accompanied by a caregiver who can assist with study procedures, provide demographic and experience-related information, and record brief home activity videos.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-10-22 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Virtual Upper-Limb Assessments: Completion Rate of Virtual aROM | From enrollment through completion of the 2 virtual assessments (approximately 2 weeks).
  The percentage of enrolled participants who complete the virtually administered active range of motion (aROM) assessment. Feasibility success is defined a priori as >70% completion.
Feasibility of Virtual Upper-Limb Assessments: Completion Rate of Virtual Box and Block Test (BBT) | From enrollment through completion of the 2 virtual assessments (approximately 2 weeks).
  The percentage of enrolled participants who complete the virtually administered Box and Block Test (BBT). Feasibility success is defined a priori as >70% completion.
Feasibility of Virtual Upper-Limb Assessments: Completion Rate of Virtual Quality of Upper Extremity Skills Test (QUEST) | From enrollment through completion of the 2 virtual assessments (approximately 2 weeks).
  The percentage of enrolled participants who complete the virtually administered Quality of Upper Extremity Skills Test (QUEST). Feasibility success is defined a priori as >70% completion.
Feasibility of Virtual Upper-Limb Assessments: Completion Rate of Virtual SHUEE Spontaneous Functional Analysis (SHUEE-SFA) | From enrollment through completion of the 2 virtual assessments (approximately 2 weeks).
  The percentage of enrolled participants who complete the virtually administered SHUEE Spontaneous Functional Analysis (SHUEE-SFA). Feasibility success is defined a priori as >70% completion.
Feasibility of Virtual Upper-Limb Assessments: Recruitment and Attrition Metrics | From enrollment through completion of participation (approximately 3-4 weeks).
  Recruitment rate (number of participants enrolled over the recruitment period), attrition rate (percentage of enrolled participants who do not complete the virtual assessment component), and documented reasons for non-eligibility, non-participation, or withdrawal.
Feasibility of Virtual Upper-Limb Assessments: Ability to Obtain Required Household Materials for Virtual Assessment | Prior to commencement of virtual assessments (Week 1)
  The percentage of families who report successfully obtaining all required household materials needed to complete the virtual standardized assessments from home.
Feasibility of Virtual Upper-Limb Assessments: Technical, Environmental, Behavioral, and Cognitive Challenges During Virtual Sessions | During Virtual Assessment 1 and Virtual Assessment 2 (approximately 2 weeks)
  The number of technical (e.g., dropped connection), video quality (e.g., lighting, camera angle), behavioral (e.g., distraction), and cognitive (e.g., confusion) challenges observed during virtual assessment sessions, coded from session videos using the standardized Observational Checklist and Behavioural Observation Research Interactive Software (BORIS).
Feasibility of Virtual Upper-Limb Assessments: Duration of Virtual and In-Person aROM | During Virtual Assessment #1, Virtual Assessment #2 and In-Person Assessment Session #1 (approximately 3 weeks)
  Time required to complete the active range of motion (aROM) when administered virtually compared to in person, as recorded using the standardized Observational Checklist.
Feasibility of Virtual Upper-Limb Assessments: Duration of Virtual and In-Person BBT | During Virtual Assessment #1, Virtual Assessment #2 and In-Person Assessment Session #1 (approximately 3 weeks)
  Time required to complete the Box and Blocks Test (BBT) when administered virtually compared to in person, as recorded using the standardized Observational Checklist.
Feasibility of Virtual Upper-Limb Assessments: Duration of Virtual and In-Person QUEST | During Virtual Assessment #1, Virtual Assessment #2 and In-Person Assessment Session #1 (approximately 3 weeks)
  Time required to complete the QUEST when administered virtually compared to in person, as recorded using the standardized Observational Checklist.
Feasibility of Virtual Upper-Limb Assessments: Duration of Virtual and In-Person SHUEE-SFA | During Virtual Assessment #1, Virtual Assessment #2 and In-Person Assessment Session #1 (approximately 3 weeks)
  Time required to complete the SHUEE-SFA when administered virtually compared to in person, as recorded using the standardized Observational Checklist.
Acceptability of Virtual aROM (Caregiver and Therapist) | Immediately after each virtual and in-person assessment (weeks 1-3).
  Acceptability of virtual administration of the active range of motion (aROM) assessment will be measured using a post-session Acceptability Survey administered via REDCap. After each assessment session, caregivers and the occupational therapist will each rate whether the virtual administration of the aROM was comparable or preferable to in-person administration. Acceptability success is defined a priori as >70% comparable or preferable ratings.
Acceptability of Virtual Box and Block Test (Caregiver and Therapist) | Immediately after each virtual and in-person assessment (weeks 1-3).
  Acceptability of virtual administration of the Box and Block Test will be measured using a post-session Acceptability Survey administered via REDCap. After each assessment session, caregivers and the occupational therapist will each rate whether the virtual administration of the BBT was comparable or preferable to in-person administration. Acceptability success is defined a priori as >70% comparable or preferable ratings.
Acceptability of Virtual QUEST (Caregiver and Therapist) | Immediately after each virtual and in-person assessment (weeks 1-3).
  Acceptability of virtual administration of the QUEST will be measured using a post-session Acceptability Survey administered via REDCap. After each assessment session, caregivers and the occupational therapist will each rate whether the virtual administration of the QUEST was comparable or preferable to in-person administration. Acceptability success is defined a priori as >70% comparable or preferable ratings.
Acceptability of Virtual SHUEE-SFA (Caregiver and Therapist) | Immediately after each virtual and in-person assessment (weeks 1-3).
  Acceptability of virtual administration of the SHUEE-SFA will be measured using a post-session Acceptability Survey administered via REDCap. After each assessment session, caregivers and the occupational therapist will each rate whether the virtual administration of the SHUEE-SFA was comparable or preferable to in-person administration. Acceptability success is defined a priori as >70% comparable or preferable ratings.
Equivalence of Virtual and In-Person aROM Scores | Across the two virtual assessments and subsequent in-person assessment (approximately 3 weeks).
  Agreement between virtual and in-person assessment aROM scores (scored live, 2-3 days apart) will be examined using mean absolute differences, intraclass correlation coefficients (ICCs; target ICC ≥0.90, lower 95% CI >0.60), Bland-Altman limits of agreement, and coefficient of variation (<10%). Equivalence is met if 80% confidence limits fall within each test's minimally important change or smallest detectable difference. Factors contributing to low agreement (e.g., internet quality, scope of view) will be explored using session videos.
Equivalence of Virtual and In-Person BBT Scores | Across the two virtual assessments and subsequent in-person assessment (approximately 3 weeks).
  Agreement between virtual and in-person assessment BBT scores (scored live, 2-3 days apart) will be examined using mean absolute differences, intraclass correlation coefficients (ICCs; target ICC ≥0.90, lower 95% CI >0.60), Bland-Altman limits of agreement, and coefficient of variation (<10%). Equivalence is met if 80% confidence limits fall within each test's minimally important change or smallest detectable difference. Factors contributing to low agreement (e.g., internet quality, scope of view) will be explored using session videos.
Equivalence of Virtual and In-Person QUEST Scores | Across the two virtual assessments and subsequent in-person assessment (approximately 3 weeks).
  Agreement between virtual and in-person assessment QUEST scores (scored live, 2-3 days apart) will be examined using mean absolute differences, intraclass correlation coefficients (ICCs; target ICC ≥0.90, lower 95% CI >0.60), Bland-Altman limits of agreement, and coefficient of variation (<10%). Equivalence is met if 80% confidence limits fall within each test's minimally important change or smallest detectable difference. Factors contributing to low agreement (e.g., internet quality, scope of view) will be explored using session videos.
Equivalence of Virtual and In-Person SHUEE-SFA Scores | Across the two virtual assessments and subsequent in-person assessment (approximately 3 weeks).
  Agreement between virtual and in-person assessment SHUEE-SFA scores (scored live, 2-3 days apart) will be examined using mean absolute differences, intraclass correlation coefficients (ICCs; target ICC ≥0.90, lower 95% CI >0.60), Bland-Altman limits of agreement, and coefficient of variation (<10%). Equivalence is met if 80% confidence limits fall within each test's minimally important change or smallest detectable difference. Factors contributing to low agreement (e.g., internet quality, scope of view) will be explored using session videos.
Test-Retest Reliability of Virtual aROM | Between Virtual Assessment 1 and Virtual Assessment 2 (1-week interval).
  Reliability will be evaluated using ICCs for (a) the two virtual assessments performed one week apart (live scoring), and (b) live scoring versus video-based scoring. Paired t-tests will examine systematic differences across repeated sessions.
Test-Retest Reliability of Virtual BBT | Between Virtual Assessment 1 and Virtual Assessment 2 (1-week interval).
  Reliability will be evaluated using ICCs for (a) the two virtual assessments performed one week apart (live scoring), and (b) live scoring versus video-based scoring. Paired t-tests will examine systematic differences across repeated sessions.
Test-Retest Reliability of Virtual QUEST | Between Virtual Assessment 1 and Virtual Assessment 2 (1-week interval).
  Reliability will be evaluated using ICCs for (a) the two virtual assessments performed one week apart (live scoring), and (b) live scoring versus video-based scoring. Paired t-tests will examine systematic differences across repeated sessions.
Test-Retest Reliability of Virtual SHUEE-SFA | Between Virtual Assessment 1 and Virtual Assessment 2 (1-week interval).
  Reliability will be evaluated using ICCs for (a) the two virtual assessments performed one week apart (live scoring), and (b) live scoring versus video-based scoring. Paired t-tests will examine systematic differences across repeated sessions.
Predictors of Feasibility, Acceptability, and Equivalence | From enrollment through completion of participation (approximately 3-4 weeks).
  Logistic regression analyses will examine whether participant characteristics (age, disability level [MACS], gender, sex, ethnicity, socioeconomic status) predict three dichotomized outcomes: (1) completion of virtual standardized assessments (yes/no), (2) willingness to participate in future virtual assessments (yes/no), and (3) acceptable agreement between virtual and in-person assessment scores (yes/no).

SECONDARY OUTCOMES:
Feasibility of Caregiver-Recorded Activity Videos (PQRS) | During weeks 1-3.
  Proportion of families who successfully produce two scorable activity videos following (a) in-person therapist instruction and (b) virtual therapist instruction. Success defined as >70% scorable videos.
Acceptability of Caregiver-Recorded Videos | Immediately after video submission (weeks 1-3).
  Percentage of families reporting satisfaction with video recording as a component of assessment, using an a priori threshold of >70% satisfaction.
Test-Retest Reliability of Perceived Quality Rating Scale (PQRS) Scores | Across two video-recording periods separated by approximately 1 week
  Test-retest reliability of caregiver-recorded activity videos will be evaluated using intraclass correlation coefficients (ICCs), a unitless reliability statistic, calculated across two sets of videos recorded approximately one week apart for the same individualized activities and scored using the Perceived Quality Rating Scale (PQRS).
Feasibility of Gamified Assessment Tasks | During the in-person assessment (week 3).
  Percentage of participants who successfully complete all gamified tasks.
Acceptability of Gamified Assessment Tasks | In-person assessment (Week 3).
  Measured by the caregiver using a post-session Acceptability Survey administered via REDCap following the in-person assessment session.
Convergent Validity of Gamified Movement Metrics | During in-person assessment (week 3).
  Correlations will be computed between kinematic outputs (e.g., smoothness, peak velocity, reach envelope, symmetry) and established clinical assessments (e.g., aROM, AHA symmetry scores).
Feasibility of Wrist-Worn Inertial Sensors | 5-day home monitoring period (week 2).
  Percentage of participants who successfully collect >15 hours of usable sensor data over 5 days, and the proportion who wear sensors during in-person assessment when appropriate.
Acceptability of Inertial Sensors | Immediately after sensor-wear period (week 2).
  Measured as the percentage of children who report willingness to wear the sensors again following completion of the sensor wear period.
Convergent Validity of Inertial Sensor Activity Counts | During the 5-day sensor-wear period and in-person assessment session (weeks 2-3).
  Assessed using correlation analyses between SHUEE Spontaneous Functional Analysis (SHUEE-SFA) scores and acceleration-derived activity counts and activity-count ratios for the dominant and hemiplegic limb. Activity counts will be derived using (i) an established threshold-based method and (ii) a machine-learning-based classifier, with activity counts from the best-performing classifier used in the correlation analysis.
Performance of Machine-Learning Classifier for Functional Arm Use | During data analysis following completion of inertial sensor data collection
  Performance of the machine-learning classifier used to classify functional and non-functional arm movements will be evaluated using precision, recall, and F1-score, based on Leave-One-Subject-Out cross-validation.

OTHER OUTCOMES:
Qualitative Themes on Experiences With Virtual and In-Person Assessment | Week 4
  Semi-structured interviews with children, caregivers, and therapists will be analyzed using reflexive thematic analysis. Outcomes include themes and subthemes describing perceptions of feasibility, acceptability, barriers, facilitators, and recommendations for implementation.
Integrated Mixed-Methods Findings on Feasibility, Acceptability, Equivalence and and Family/Clinician Experience | After completion of all quantitative and qualitative analyses (approximately weeks 4-6 following the final participant visit)
  Quantitative and qualitative data will be merged following their initial analyses to examine complementarity, convergence, and divergence, as well as family and clinician experiences with virtual and in-person assessments. Integration will use a weaving approach, with qualitative and quantitative findings presented together by theme and summarized narratively and through joint displays. Side-by-side joint displays will compare quantitative indicators (e.g., demographics, number of technical issues) with qualitative data (e.g., interview quotes) to contextualize preferences and experiences related to virtual and in-person assessment. Joint displays will organize qualitative themes by Theoretical Domains Framework (TDF) domains to support interpretation of clinician and family experiences.

CONTACTS AND LOCATIONS:
Overall Officials: Elaine Biddiss, PhD, Principal Investigator — Holland Bloorview Kids Rehabilitation Hospital, Bloorview Research Institute; Virginia Wright, PhD, Principal Investigator — Holland Bloorview Kids Rehabilitation Hospital, Bloorview Research Institute
Locations (3):
- Canada (3):
  - Grandview Kids, Ajax, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Holland Bloorview Kids Rehabilitation Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No